CLINICAL TRIAL: NCT03334682
Title: Randomized Double-blind Study on the Benefit of Spironolactone for Treating Acne of Adult Woman.
Acronym: FASCE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RC16_0467
Record Dates: First submitted 2017-10-30; First posted 2017-11-07 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Spironolactone; Doxycycline

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The products used in both arms will be over-encapsulated by the Pharmacy of Nantes University Hospital
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- spironolactone (Experimental): Spironolactone ARROW ® 75 mg, 150mg, orally, once a day during all the trial (12 months: 6 months on double-blinded spironolactone then 6 months on open-label spironolactone), + topical therapy during all the trial (benzoyl peroxide 5%)
  Interventions: Drug: spironolactone
- doxycycline (Active Comparator): (Doxycycline Sandoz 100 mg), 100mg/day during 3 months followed by placebo during 3 months, on double-blinded + topical therapy during all the trial (benzoyl peroxide 5%
  Interventions: Drug: Doxycycline

INTERVENTIONS:
Drug: spironolactone — Dispensation of spironolactone at each visit according to the arm description described above.
  Arms: spironolactone
Drug: Doxycycline — Dispensation of doxycycline then placebo, at each visit according to the arm description described above.
  Arms: doxycycline

SUMMARY:
Acne vulgaris of adult woman has increased over the past 10 years; it affects currently 20% to 30% of adult women.

The physiopathology of adult woman acne is distinguished from the teenager one by essentially 2 factors:

* hormonal factor with a peripheral hyperandrogenism coupled with an hypersensibility of cutaneous androgens receptors of these women. But this point is still at the stage of hypothesis.
* inflammatory factor linked with Propionibacterium Aces ; indeed these women received most of the time many cures of local and systematic antibiotics at the origin of resistant Propionibacterium Aces strains which lead to a chronical activation of cutaneous innate immunity.

On a therapeutic plan, four types of systemic treatment, approved in this indication are:

* Tetracyclines which are problematic for the bacterial resistance and consequently constant relapse when they are stopped.
* Zinc salts which target only the inflammatory lesions and were shown less effective than cycline
* Antiandrogens, with acetate of cyproterone associated with risks of phlebitis and pulmonary embolism, and increase risk of triglycerides, cholesterol and hepatic balance.
* The last alternative is represented by isotretinoin but the use in women of childbearing potential is binding because of the teratogen risks and the hyperandrogenism represents an identified risk of relapse.

In this context, the spironolactone could represent an interesting alternative. It blocks the 5-alpha-reductase receptors at sebaceous gland and inhibits Luteinizing hormone (LH) production at the pituitary level. It is not submitted to isotretinoin constraints, does not lead to bacterial resistance and targets the peripheral hyperandrogenism.

Currently, very few studies have been performed and on a weak number of patients but they showed that at low doses (lower than 200mg/day), spironolactone can be effective against acne.

In that context, it seemed clearly interesting to perform the first double-blind randomized study spironolactone vs cyclines which remains the moderate acne reference treatment and to demonstrate the superiority of spironolactone's efficacy in order to establish it as alternative way to cycline.

ELIGIBILITY:
Inclusion Criteria:

* Patient with acne, with at least 10 inflammatory lesions and no more than 3 nodules
* Patient who already had one cycline course for her acne treatment with a 3 months* wash out or who never had any cycline
* Patient having signed an informed consent
* Absence of use of oral antibiotics and Zinc salts in the last 30 days
* Absence of use of systemic isotretinoin and antiandrogens in the last 6 months
* Absence of microphysiotherapy in the last 15 da
* Women of child-bearing age under contraception since 3 months (oral contraception, implant or IUD).
* Patients with social security

Exclusion Criteria:

* Patient affected by active /progressive diseases, as infections including Hidradenitis suppurativa, cancers, or endocrine syndrome (eg polycystic ovary syndrome), Addison's disease)
* Patient affected by Rosacea
* Patient with contra-indication to the use of one of the investigational products or auxiliary :

  * Patient with intolerance or hypersensitivity to cyclin's, spironolactone or to any ingredient present in associated benzoyl peroxide gel
  * Patient with significant impairment of renal excretory function, acute or chronic renal failure, anuria.
  * Patient with life-threatening or very severe hepatic impairment.(grade III or IV)
* Patient with hyperkalaemia or strongly requiring potassium-sparing diuretics (eg amiloride, canrenoate, eplerenone, triamterene), or treated continuously with Angiotensin-converting-enzyme (ACE) inhibitors, angiotensin II antagonist, NSAIDs, heparin and molecular weight heparin, ciclosporin and tacrolimus.
* Patient requiring topical isotretinoin or who stopped this drug since less than 2 weeks
* Patient previously treated with spironolactone
* Pregnant woman or likely to become pregnant or nursing and refusing to use an effective contraceptive method
* Patient participating in another interventional clinical trial
* Patient under guardianship or trusteeship

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2023-02-03 (Actual); Study Completion 2023-07-04 (Actual)

PRIMARY OUTCOMES:
Treatment efficacy | Month 4 and Month 6
  The treatment's efficacy will be determined by the rate of success in each arm. The best rate of success between Month 4 and Month 6 will be chosen for the final result. Rate of success, defined by a decrease of both Adult Female Acne Scoring Tool (AFAST) scores 1 and 2:
  1. AFAST score 1: decrease of at least 2 grades compared to baseline or to grade 0 if the baseline was at 1 and
  2. AFAST score 2: decrease to grade 1 if baseline was > 1 or to grade 0 if the baseline was at 1
  AFAST 1 (also called GEA) assesses the comedones (open and closed), the non-inflammatory lesions, the papules and pustules and the nodules. The stage is defined according to a global evaluation of severity of acne and ranges from Grade 0 (no acne) to Grade 5 (the worse situation).
  AFAST 2 assesses acne on an area from the left and right mandibular zone to the upper edge of the trunk and ranges from Grade 0 (no acne) to Grade 3 (the worse situation).

SECONDARY OUTCOMES:
Clinical adverse events | Within 12 months after randomization
  Number and type of Adverse Events (AE) and Serious Adverse Events (SAE) occurring from the beginning of the treatment until end of the follow-up
Sodium abnormal values (biological adverse events) | From 30 days to 7 days before randomization visit, Month 2, Month 4, Month 9
  Sodium measurement (mmol/L)
Potassium abnormal values (biological adverse events) | From 30 days to 7 days before randomization visit, Month 2, Month 4, Month 9
  potassium measurement (mmol/L)
Chlore abnormal values (biological adverse events) | From 30 days to 7 days before randomization visit, Month 2, Month 4, Month 9
  Chlore measurement (mmol/L)
Calcium abnormal values (biological adverse events) | From 30 days to 7 days before randomization visit, Month 2, Month 4, Month 9
  Calcium measurement (mmol/L)
AFAST score 1 (GEA) at 0 or 1 | Month 2, Month 4, Month 6, Month 9 and Month 12
  Number of patients with AFAST score 1 (GEA) at 0 or 1.
AFAST score 2 (Mandibular) at 0 or 1 | Month 2, Month 4, Month 6, Month 9 and Month 12
  Number of patients with AFAST score 2 (Mandibular) at 0 or 1.
AFAST score 1 associated with AFAST score 2 at 0 or 1 | M2, M4, M6, M9 and M12
  Number of patients with both AFAST score 1 and AFAST score 2 at 0 or 1.
Quality of life (cost-utility assessment and general quality of life assessment) | Month 2, Month 4, Month 6, Month 9 and Month 12
  EQ-5D (EuroQol 5 dimensions) questionnaire: The questionnaire focuses on five dimensions: mobility, personal autonomy, current activities, pain/discomfort, and anxiety/depression. For each of these dimensions, three answers are possible.
Quality of life (specific to acne) | Month 2, Month 4, Month 6, Month 9 and Month 12
  Cardiff Acne disability Index (CADI) is a disease-specific questionnaire measuring disability induced by acne.
Bacterial and parasital evaluations | Day 0 (baseline) and Month 4
  Presence of P acnes, M Furfur and S epidermidis, aureus
Inflammatory lesions of the face | Day 0 (baseline), Month 2, Month 4, Month 6, Month 9 and Month 12
  Number of inflammatory lesions of the face
retentional lesions of the face | Day 0 (baseline), Month 2, Month 4, Month 6, Month 9 and Month 12
  Number of retentional lesions of the face
Face lesions | Day 0 (baseline), Month 2, Month 4, Month 6, Month 9 and Month 12
  Total number of face lesions
Trunk lesions | Day 0 (baseline), Month 2, Month 4, Month 6, Month 9 and Month 12
  Factor F2 of ECLA scale ECLA ("Echelle de Cotation des Lésions d'Acné") is a scale for acne proposed by the dermatology research team of Nantes University Hospital. It is composed of 3 factors: Factor 1 (F1) counts the acne lesions on the face; Factor 2 (F2) counts the lesions acne on the trunk and Factor 3 (F3) counts the scars. In this study, the factor F2 will be used. The factor F2 assesses the extensive character of acne lesions on 5 defined areas: cervical areas (F2N); chest areas (F2C); back area (F2B) and arm area (F2A) according to a qualitative scale 0=absent, 1=poor 2=medium 3=significant. It is completed by the count of the present nodules in each area.
Relapse | Month 4 and Month 6
  number of patients with relapse, defined as follows :
  1. AFAST score 1 (GEA score): increase of 2 points versus score of previous visit, in case of success Or
  2. AFAST score 2 (mandibular score): increase of 1 point versus score of previous visit, in case of success
Reappearance of 10% and more of inflammatory lesions. | Month 6
  Number of patients with a reappearance of 10% and more of inflammatory lesions.
Incremental cost-effectiveness ratio (cost per Quality-Adjusted Life-Year, QALY) of the comparison between the spironolactone and cycline. | Month 6
  costs: resources consumed, QALY: EQ-5D

CONTACTS AND LOCATIONS:
Locations (9):
- France (9):
  - Chru Brest, Brest
  - CHU Caen, Caen
  - CHU Grenoble, Grenoble
  - CH La Rochelle, La Rochelle
  - CH Le Mans, Le Mans
  - CHU de Nantes - Dermatologie, Nantes
  - CHU Poitiers, Poitiers
  - Cabinet du Dr Jean-Paul Claudel, Tours
  - CHRU Tours, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Poinas A, Lemoigne M, Le Naour S, Nguyen JM, Schirr-Bonnans S, Riche VP, Vrignaud F, Machet L, Claudel JP, Leccia MT, Hainaut E, Beneton N, Dert C, Boisrobert A, Flet L, Chiffoleau A, Corvec S, Khammari A, Dreno B. FASCE, the benefit of spironolactone for treating acne in women: study protocol for a randomized double-blind trial. Trials. 2020 Jun 25;21(1):571. doi: 10.1186/s13063-020-04432-w. PMID 32586344